CLINICAL TRIAL: NCT05881733
Title: Effect of a Bigger Cryoballoon on the Total Antral Lesion Size: Evaluation of POLARx FIT
Acronym: BETTER-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Sing-Chien Yap, MD, PhD, Cardiologist-electrophysiologist, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2023-0325; NL84423.078.23 (Registry Identifier: CCMO)
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
Keywords: Cryoballoon; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, single-center, study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Other): This study will have only a single arm. Patients will undergo pulmonary vein isolation using the 31 mm balloon size of POLARx FIT. High-definition 3D maps will be constructed before and after cryoablation to assess the antral lesion size.
  Interventions: Device: POLARx FIT cryoballoon

INTERVENTIONS:
Device: POLARx FIT cryoballoon — Patients will undergo cryoablation with the 31 mm balloon size of the POLARx FIT cryoballoon.

SUMMARY:
The investigators will prospectively evaluate the extent of antral lesion created by the 31 mm balloon size of a novel cryoballoon catheter (POLARx FIT). In 20 patients with paroxysmal atrial fibrillation, the investigators will perform pre- and post-ablation high-definition 3D maps to quantify the extent of lesion created by the 31 mm POLARx FIT cryoballoon.

DETAILED DESCRIPTION:
Rationale: The next generation POLARx cryoablation balloon (CB) catheter will have the option of to deliver cryotherapy with the current balloon size of 28 mm or a new, larger 31 mm size by changing the inner balloon pressure (POLARx FIT, Boston Scientific). Currently, there is no data on the extension of left atrial (LA) lesion formation with the 31 mm balloon size of the POLARx FIT cryoablation balloon catheter. The hypothesis is that a larger CB size results in a wide antral circumferential lesion.

Objective: The primary objective is to evaluate the antral lesion size using ultrahigh-density (UHDx) mapping pre- and post-cryoablation with the 31 mm balloon size CB. Secondary objectives are the proportion of pulmonary veins (PVs) where a 31 mm CB could be positioned to achieve a grade 4 occlusion and the single shot success rate with the 31 mm balloon size CB.

Study design: Single-center, single-arm, prospective study with pre- and post-PVI UHDx mapping.

Study population: Twenty adult patients with paroxysmal AF who are scheduled to undergo pulmonary vein isolation (PVI) with a CB.

Intervention: Patients will undergo pre- and post-ablation UHDx mapping (Orion catheter and Rhythmia 3D-mapping system, Boston Scientific) during the index procedure.

Main study parameters/endpoints: The primary endpoint is the extent of the antral lesion size. Secondary endpoints are the proportion of PVs with grade 4 occlusion with the 31 mm balloon size CB, the single shot success rate of the 31 mm balloon size CB, difference in rate of achieving grade 4 occlusion in comparison to the standard (28 mm) size.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: A UHDx mapping will be acquired before and after complete PVI. The procedures will be performed under deep sedation, which is standard practice for CB procedures in our institution. The risk of additional mapping is limited. LA mapping is a standard diagnostic method for patients undergoing PVI with radiofrequency ("standard-of-care"). In the current study, UHDx mapping will now be used in patients undergoing PVI with CB. The most important complication of additional intracardiac mapping is cardiac tamponade, but this risk is low (<0.5%).

ELIGIBILITY:
Inclusion Criteria:

1. History of symptomatic paroxysmal AF
2. Subjects who are indicated for a PVI according to the 2020 ESC guidelines for the diagnosis and management of AF
3. Subjects who are willing and capable of providing informed consent
4. Subjects who are willing and capable of participating in all testing associated with this clinical investigation
5. Subjects whose age is 18 years or above

Exclusion Criteria:

1. Any known contraindication to an AF ablation or anticoagulation
2. History of previous left atrial ablation or surgical treatment of AF, atrial flutter, or atrial tachycardia
3. AF secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause
4. Significant structural heart disease as evidenced by:

   1. Left ventricular ejection fraction <45% based on most recent transthoracic echocardiogram (TTE) performed <6 months prior to enrollment
   2. LA diameter >55 mm based on most recent TTE performed <6 months prior to enrollment
   3. Previous cardiac surgery
   4. Previous cardiac valvular surgical or percutaneous procedure
   5. Interatrial baffle, closure device, patch, or occluder
   6. Unstable angina or ongoing myocardial ischemia
   7. Moderate or severe valvular heart disease on most recent TTE performed <6 months prior to enrolment
   8. Congenital heart disease
   9. Left atrial thrombus
5. History of blood clotting or bleeding disease
6. Stroke or transient ischemic attack <3 months prior to enrollment
7. Active systemic infection
8. Common ostium PV >24 mm defined by CT-scan
9. Pregnant, lactating, or women of childbearing potential who are, or plan to become, pregnant during the time of the study
10. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sing-Chien Yap, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study population
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Ablated Left Atrial Posterior Wall With a 31 mm Balloon Size POLARx FIT
Description: Low-voltage areas will be quantified using a bipolar voltage <0.3 mV. The sum of the posterior ablated areas of all pulmonary veins is expressed as a percentage of the total left atrial posterior wall.
Time Frame: Interprocedural (directly after cryoablation)
Measure: Mean (Standard Deviation); unit: percentage of posterior wall
Arm/Group | Study population
Number analyzed (Participants) | 20
percentage of posterior wall | 35.4 (13.8)

2. Secondary Outcome: Percentage of Pulmonary Veins With Grade 4 Occlusion With a 31 mm Balloon Size POLARx FIT
Description: A grade 4 occlusion is defined as complete contrast stasis. Cine acquisitions of contrast vein occlusions was analyzed by two experienced observers.
Time Frame: Interprocedural (before cryoablation)
Population: There were 4 pulmonary veins per participant. Thus, in 20 participants there were 80 pulmonary veins. We determined the percentage of pulmonary veins which had a grade 4 occlusion with the 31 mm balloon size of the POLARx FIT catheter. In 69 of 80 pulmonary veins (86%) a grade 4 occlusion with the 31 mm balloon size could be achieved.
Measure: Number; unit: Percentage
Units Other Than Participants: Pulmonary_veins
Arm/Group | Study population
Number analyzed (Participants) | 20
Number analyzed (Pulmonary_veins) | 80
Percentage | 86

3. Secondary Outcome: Percentage of Pulmonary Veins With a Single Shot Success Rate Using a 31 mm Balloon Size POLARx FIT Cryoablation Catheter
Description: Pulmonary vein isolation will be determined using conventional criteria: entry- and exit-block as assessed with the circular mapping catheter (POLARMAP).
Time Frame: Interprocedural (directly after cryoablation)
Population: There were 4 pulmonary veins per participant. Thus, in 20 participants there were 80 pulmonary veins. We determined the percentage of pulmonary veins which were isolated after 1 cryoapplication with the 31 mm balloon size of the POLARx FIT catheter. 63 of 80 pulmonary veins (79%) were isolated after 1 cryoapplication.
Measure: Number; unit: Percentage
Units Other Than Participants: Pulmonary_veins
Arm/Group | Study population
Number analyzed (Participants) | 20
Number analyzed (Pulmonary_veins) | 80
Percentage | 79

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Study population
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study population (N=20)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) — Esophageal perforation requiring major surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT05881733/Prot_SAP_000.pdf